CLINICAL TRIAL: NCT06210568
Title: Role of Oxidative Stress in Male Infertility: an Observational Case-control Study
Brief Title: Oxidative Stress and Male Infertility.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Enrico Papaleo, MD, IRCCS San Raffaele
Other Study IDs: INAIL OSES2022
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infertile Male Patients
  Interventions: Other: no intervention
- Fertile males
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Study Aims:

To evaluate the impact of oxidative and nitrosative stress, as well as DNA methylation, on male reproductive health. This is achieved by analyzing urinary biomarkers: 8-oxoGua, 8-oxoGuo, 8-oxodGuo, 3-nitrotyrosine (3-NO2Tyr), 5-methylcytidine (5-MeCyt), and cotinine in infertile and fertile males.

Study Design:

A prospective observational case-control study comparing infertile male patients (cases) from a reproductive sciences center with fertile male volunteers (controls) from a gynecology and obstetrics department. The study focuses on understanding the role of oxidative stress in male infertility and its implications for assisted reproductive techniques.

DETAILED DESCRIPTION:
Infertility affects approximately 15% of couples in their reproductive age. Male factors contribute to 45-50% of infertility cases, with 7% of the global male population diagnosed as infertile. Oxidative stress, defined as an imbalance between reactive oxygen species (ROS) and antioxidants, plays a significant role in semen quality degradation. High levels of ROS, unbalanced by antioxidant mechanisms, damage spermatozoa, affecting motility and morphology, and compromising their fertilizing ability. Excessive ROS production, antioxidant depletion, and inactivation or reduced production of antioxidant enzymes contribute to this imbalance. Oxidative stress not only induces lipid peroxidation in sperm membranes but also impacts DNA integrity and increases apoptosis rates. It is estimated to be a significant factor in 30-80% of male infertility cases. Oxidative and nitrosative stress are interrelated; increased ROS levels can interact with nitrogen species, causing further reproductive function damage. Urinary oxidized nucleic acid bases, particularly 8-oxo-7,8-dihydroguanine (8-oxoGua) and 8-oxo-7,8-dihydro-2'-deoxyguanosine (8-oxodGuo), serve as biomarkers of oxidative stress. Additionally, DNA methylation plays a crucial role in biological processes, with 5-methylcytidine (5-MeCyt) acting as an epigenetic biomarker.

Objectives:

The primary objective is to assess the role of oxidative, nitrosative stress, and DNA methylation on male reproductive health by evaluating urinary biomarkers: 8-oxoGua, 8-oxoGuo, 8-oxodGuo, 3-nitrotyrosine (3-NO2Tyr), 5-MeCyt, and cotinine. The secondary objectives include evaluating semen quality parameters impacted by oxidative stress and identifying potential environmental and lifestyle exposure sources contributing to oxidative stress.

Study Design:

This monocentric, prospective observational study will involve two patient groups: infertile male patients ("cases") attending the Center for Reproductive Sciences and fertile male volunteers ("controls") from the Department of Gynecology and Obstetrics. Procedures for patients and volunteers are additional to the study protocol and not experimental in nature. The study aims to provide a comprehensive understanding of oxidative stress in male infertility and its potential impact on assisted reproductive techniques.

ELIGIBILITY:
Inclusion Criteria:

Infertile Male Patients: a diagnosis of couple infertility due to no conception for over 12 months (as per the access criteria for Assisted Reproductive Technology defined by law 40/2004), aged between 18 and 50 years, and having signed informed consent.

Fertile Males:Inclusion criteria are having fathered at least one child, aged between 18 and 50 years, and having signed informed consent.

Exclusion Criteria:

Infertile Male Patients: Exclusion criteria include a clear diagnosis of infertility due to established clinical evidence (evident endocrinological disorders, previous testicular trauma, vasectomy, epididymitis, orchitis, cryptorchidism, varicocele), inability to produce a useful semen sample for analysis (azoospermia), past diseases that involved radiological therapies in the genital area, and creatinuria levels outside the WHO normal range (0.3-3 grams).

Fertile Males:conception using assisted reproductive techniques and a waiting time of more than 12 months for conception, as well as creatinuria levels outside the WHO normal range (0.3-3 grams).

Ages: 18 Years to 50 Years | Sex: Male
Age Groups: Adult
Study Population: The study includes 800 males in two groups. Group 1: 400 males from the Center for Reproductive Sciences, aged 18-50, diagnosed with infertility after over 12 months of unsuccessful conception (ART criteria, law 40/2004). Exclusions: clear infertility diagnoses (endocrinological disorders, testicular trauma, vasectomy, epididymitis, orchitis, cryptorchidism, varicocele, azoospermia), past genital radiological treatments, abnormal WHO creatinuria (0.3-3 grams).
  Group 2: 400 healthy males from Obstetrics and Gynecology, aged 18-50, who fathered a child naturally within 12 months. Exclusions: ART conception, over 12 months for conception, abnormal WHO creatinuria levels.
  This diverse population enables analyzing oxidative stress's role in male infertility, comparing infertile and fertile males' biological markers and health profiles.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of oxidative and nitrosative stress, as well as DNA methylation, on male reproductive health. | 2 years
  Analyze urinary biomarkers: 8-oxoGua, 8-oxoGuo, 8-oxodGuo, 3-nitrotyrosine (3-NO2Tyr), 5-methylcytidine (5-MeCyt), and cotinine in infertile and fertile males.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Papaleo, Study Director — IRCCS San Raffaele; Luca Pagliardini, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No